CLINICAL TRIAL: NCT04103190
Title: Multiparametric Imaging for Analysis of MVNT (Multinodular and Vacuolating Neuronal Tumor)
Acronym: MIAM
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: ALR_2019_4
Record Dates: First submitted 2019-06-21; First posted 2019-09-25 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Benign Neuronal Desease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: cerebral MRI — Patients who agree to participate in the study will perform a 3T multi-parametric MRI with advanced spectroscopic imaging techniques and standard protocol.
  A neurological consultation will take place during the inclusion visit as well as a questionnaire and a control MRI at 1 year and 2 years +/- 1 month.

SUMMARY:
Differential diagnoses of MVNT include DNT (dysembryoplastic neuroepithelial tumor), low-grade gliomas, cortical dysplasias or even hamartomas.

DETAILED DESCRIPTION:
Differential diagnoses of MVNT include DNT (dysembryoplastic neuroepithelial tumor), low-grade gliomas, cortical dysplasias or even hamartomas.

However, in order to avoid an invasive surgical procedure to remove the lesion, a certain diagnosis of its benignity is essential. The contribution of advanced techniques in MRI, such as spectroscopy in the characterization of these lesions, has not yet been studied today

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Suspicion of MVNT on an MRI: it is considered that it will be necessary at least the 2 major criteria associated with at least 1 minor criterion to enter the definition of suspicion of MVNT:

Major criteria:

* Multinodular aspect in cluster
* High FLAIR hypersignal / T2

Minor criteria:

* Absence of mass effect
* Hyposignal T1
* Center of the lesion in hypsignal FLAIR or T1 hypersignal

  * Affiliate or beneficiary of a Social Security scheme
  * Having received informed information about the study and consenting to participate in the study

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant or lactating woman
* Contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient supported for suspicion of MVNT
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Description of a new radiological entity on Spectroscopy : the MVNT (Multinodular and Vacuolating Neuronal Tumor) | 1 day
  ratio of N-Acetylaspartate / Choline on Spectroscopy
Description of a new radiological entity on Spectroscopy : the MVNT (Multinodular and Vacuolating Neuronal Tumor) | 1 day
  area under curve of the N-Acetylaspartate Spectroscopie
Description of a new radiological entity on Spectroscopy : : the MVNT (Multinodular and Vacuolating Neuronal Tumor) | 1 day
  area under curve of choline Spectroscopie

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Groupe Hospitalier Pellegrin, Bordeaux, Bordeaux
  - Fondation Adolphe de Rothschild, Paris, PARIS
  - CHU Rennes, Rennes, Rennes
  - CHU de Rouen, Rouen, Rouen
  - Hôpital Pierre Paul Riquet, CHU Purpan, Toulouse, Toulouse
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Laennec, Saint-Herblain